CLINICAL TRIAL: NCT03298217
Title: Peak Tidal Inspiratory Flow in Infants With Moderate to Severe Acute Viral Bronchiolitis: a Physiologic Study
Brief Title: Peak Tidal Inspiratory Flow in Infants With Moderate to Severe Acute Viral Bronchiolitis
Acronym: DEBIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UF9868
Record Dates: First submitted 2017-07-19; First posted 2017-10-02 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Bronchiolitis
Keywords: Inspiratory flow; High flow nasal cannula, spirometry; spirometry; physiologic study; Bronchiolitis patients sverity score mWCAS/ 3-5.
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchiolitis patients sverity (Other): In patients with bronchiolitis mWCAS / 3-5 : Measurement of the peak tidal inspiratory flow (PTIF)
  Interventions: Device: Measurement of the peak tidal inspiratory flow (PTIF)

INTERVENTIONS:
Device: Measurement of the peak tidal inspiratory flow (PTIF) — In patients with bronchiolitis sverity mWCAS / 3-5 :
  Nasopharyngeal aspiration and comfortable placement of the infant upon admission; Clinical evaluation: respiratory rate, respiratory distress scores rating (Silverman and m-WCAS); If the patient is eligible: information and collection of parental consent; If signed parental consent obtained: progressive (on at least 10 min) withdrawal of HFNC support and maintenance if necessary of conventional oxygen therapy (maximum 1 L/min); Application of the spirometer for the recording of 20 consecutive spontaneous respiratory cycles for PTIF measurements; Respiratory support with HFNC; flow adapted to the need of the patients (equal to the measured PTIF).

SUMMARY:
This aim of this study is to measure the peak tidal inspiratory flow (PTIF), using spirometry, in young infants with moderate to severe acute viral bronchiolitis (AVB).

PTIF is important to consider for the management of AVB with High Flow Nasal Cannulae (HFNC). Indeed, efficiency with HFNC is optimal provided that the settled flow is equal or higher than the patient's PTIF. However, PTIF values in infants with AVB have never been determined.

DETAILED DESCRIPTION:
HFNC allows the administration of a heated and humidified mixture of air and oxygen at high flows. This device has been widely adopted in pediatric intensive care units (PICUs) and for interhospital transport of critically ill children, as the system is easily set up and is well tolerated by patients. In the context of AVB, retrospective audits and observational studies have suggested promising outcomes on both physiological and clinical variables. However, in less than 6 months old infants with moderate to severe AVB, the failure rate with this device - defined as worsening of respiratory failure or the occurrence of discomfort or severe apnea - remains high, from 30% to 50% in key studies.

HFNC flow setting remains empiric, 2 L/kg/min being used by most teams. A potential explanation for this high failure rate is that the flow usually used is lower than the patient's inspiratory flow. The aim of this study is to determine peak tidal inspiratory flow (PTIF) values in infants up to 6 months old with moderate to severe AVB.

PTIF will be evaluated with a spirometer connected to a face mask during 20 cycles of spontaneous ventilation. The measurements will be performed within the first 24 hours of hospitalization in the department of Neonatal and Pediatric Intensive Care of Arnaud de Villeneuve University Hospital at Montpellier (France).

Statistical analysis Relation between the DIP and Silverman score, mWCAS, RR, LOS will be expressed with parametric and non-parametric correlation coefficients according to the distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* Infants up to 6 months old, with AVB according to conventional clinical criteria;
* Admitted to the department of Neonatal and Pediatric Intensive Care at Arnaud de Villeneuve University Hospital in Montpellier (France);
* Supported with HFNC, according to the department's protocol (2 < m-WCAS < 5);
* Not requiring immediate intubation for invasive ventilation;
* Signed parental consent.

Exclusion Criteria:

* Infant with heart disease, cystic fibrosis or neuromuscular disorder;
* Infant requiring ventilatory support with nasal continuous positive pressure (nCPAP) or with HFNC and without possibility of weaning, including for a few minutes;
* Intolerance of the spirometry mask.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Measurement of peak or peak inspiration flow (PTIF=peak tidal inspiratory flow) | 1 day but within 24 hours of patient admission
  Measurement of peak or peak inspiratory flow will be performed by spirometry using a spirometer within 24 hours of patient admission. Evaluation will take place within the first 24 hours of hospitalization in the department of Neonatal and Pediatric Intensive Care among patients with moderate to severe AVB.
  Description: Application of the spirometer for the recording of 20 consecutives spontaneous respiratory cycles for PTIF (l/kg/min) measurements.
  Primary outcome: average (+/-SD) of 20 consecutives PTIF.

SECONDARY OUTCOMES:
Proportion of patients with a spontaneous PTIF higher than 2 L/kg/min | 1 day but within 24 hours of patient admission
  Proportion of patients with a spontaneous PTIF higher than 2 L/kg/min
Correlation between PTIF and Silverman score | 1 day but within 24 hours of patient admission
  Correlation between PTIF (l/kg/min) and Silverman score (0 to 10)
Correlation between PTIF and modified Wood's clinical asthma score | 1 day but within 24 hours of patient admission
  Correlation between PTIF (l/kg/min) and modified Wood's clinical asthma score(m-WCAS) (0 to 10)
  * Correlation between PTIF (l/kg/min) and respiratory rate (FR) (breath/min)
  * Correlation between PTIF (l/kg/min) and carbon dioxide (CO2) (mmHg) measured by capillary blood gases or with transcutaneous electrodes, duration of hospitalization
Correlation between PTIF and respiratory rate (FR) | 1 day but within 24 hours of patient admission
  Correlation between PTIF (l/kg/min) and respiratory rate (FR) (breath/min)
Correlation between PTIF and carbon dioxide (CO2) | 1 day
  Correlation between PTIF (l/kg/min) and carbon dioxide (CO2) (mmHg) measured by capillary blood gases or with transcutaneous electrodes
Duration of hospitalization | 1 day at the end of the hospitalization
  Duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MILESI, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC